CLINICAL TRIAL: NCT05955378
Title: Assessment of a Microprocessor Ankle for Low Mobility Individuals
Brief Title: Assessing the DSR Ankle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Synchro Motion LLC (Industry)
Collaborators: Shirley Ryan AbilityLab (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STU00217993
Record Dates: First submitted 2023-07-03; First posted 2023-07-21 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Amputation; Limb Deficiencies
Keywords: Amputation; Transtibial; K2; Limited Community Ambulator

STUDY DESIGN:
Intervention Model Description: AB/BA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DSR Ankle (Experimental): The DSR Ankle is a novel microprocessor-controlled ankle prosthesis that is able to provide enhanced mobility and stability to individuals with lower limb amputation. It interfaces to the user by attaching to their socket via an industry-standard pyramid connector.
  Interventions: Device: DSR Ankle
- Predicate Ankle (Active Comparator): The predicate ankle is the user's prescribed prosthesis worn for the activities of daily living.
  Interventions: Device: Predicate Ankle

INTERVENTIONS:
Device: DSR Ankle — This is the experimental ankle component used in the overall prosthetic intervention.
  Other Names: The Damping, Stiffness and Repositioning Ankle
  Arms: DSR Ankle
Device: Predicate Ankle — This is the participant's prescribed ankle/foot complex used in the overall prosthetic intervention.
  Other Names: Daily Use Ankle
  Arms: Predicate Ankle

SUMMARY:
This research is being done to conduct a preliminary investigation into a new prosthetic microprocessor controlled (MPC) ankle, called the Damping, Stiffness, and Repositioning (DSR) ankle. The DSR ankle is a new design to support a person while they walk on both even and uneven ground, as well as with bending the ankle for safe foot clearance while a person takes a step. In particular, in this study we are interested in seeing how this type of new device may benefit people who are rated as a K2-level ambulator.

DETAILED DESCRIPTION:
Synchro Motion, LLC developed a novel MPC ankle. Because of its unique actuation scheme, the prosthesis can behave as: (1) a lockable conformal damper, (2) a variable set-point spring, and (3) an actively repositionable joint.

The investigators therefore refer to the device as the damping, stiffness, and repositioning (DSR) ankle. The DSR ankle is small, lightweight, quiet, and runs for multiple days on a single charge. No other commercially available prosthesis combines this set of features. It will be shown in preliminary work that the features of the DSR ankle can increase toe clearance in swing, reduce the time-to-foot-flat after heel strike, and improve weight bearing symmetry when standing on slopes for K3 Individuals with Lower Limb Amputation (ILLAs). These biomechanical functions have all been linked to improved safety and stability, which leads the investigators to hypothesize that the DSR ankle may provide benefits to K2 ILLAs as well.

The main purpose of this research is to determine the ways in which the DSR ankle may be adapted to provide benefits specifically to ILLAs who use their prosthesis at the K2 level. For purposes of the Phase I work, the development and assessment will be performed exclusively with K2 ILLAs in order to provide an opportunity to implement any necessary refinements to the DSR ankle to ensure optimal K2 performance. The remainder of the research is to quantify the effectiveness of the DSR ankle as compared to a predicate non-MPC ankle in improving performance for K2 ILLAs.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-89 years
2. Patients who have a unilateral transtibial amputation who are able to use a prosthesis and who currently use a passive, non-MPC prosthesis
3. K2 level ambulators

Exclusion Criteria:

1. Pregnant women
2. Children (<18 years old)
3. Prisoners or institutionalized individuals
4. Individuals who have the inability to give informed consent
5. Participants unable to walk for 2 minutes without an assistive device
6. Participants with complicating health conditions that interfere with the study
7. Inability to read and understand the English language. As this is a pilot study with a small sample size, it is prohibitive to translate Study documents to other languages as recruitment will be from a sample of convenience.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-12-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 patients were enrolled between August 22, 2023 and November 19, 2024 at the Shirley Ryan AbilityLab in Chicago, IL.
Pre-assignment Details: 3 of 5 patients completed this cross-over study.
Groups:
- Predicate Ankle, Then DSR Ankle: Participants first performed assessments with their predicate (daily use) prosthetic ankle. After a washout period of at least 2 weeks, they were trained and assessed with the DSR Ankle. The DSR Ankle is a novel microprocessor-controlled ankle prosthesis that is able to provide enhanced mobility and stability to individuals with lower limb amputation.
- DSR Ankle, Then Predicate Ankle: Participants first performed assessments with the DSR Ankle. The DSR Ankle is a novel microprocessor-controlled ankle prosthesis that is able to provide enhanced mobility and stability to individuals with lower limb amputation. After a washout period of at least 2 weeks, they were trained and assessed with their predicate (daily use) prosthetic ankle.
Period: Overall Study
Arm/Group | Predicate Ankle, Then DSR Ankle | DSR Ankle, Then Predicate Ankle
Started | 2 | 3
Completed | 2 | 1
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Predicate Ankle, Then DSR Ankle | DSR Ankle, Then Predicate Ankle | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 82 (2.8) | 59 (0) | 74.3 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Minimum Foot Clearance
Description: Minimum foot clearance is the shortest distance between the foot and the ground during swing, and it occurs approximately halfway through the swing phase of gait.
Time Frame: after up to 3 weeks of training
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | DSR Ankle | Predicate Ankle
Number analyzed (Participants) | 3 | 3
centimeters | 4.07 (0.96) | 3.87 (1.11)

2. Primary Outcome: Time to Foot Flat
Description: Time to foot flat is the duration of time between initial contact at heel strike and the full contact of the sole of the foot on the ground in stance.
Time Frame: after up to 3 weeks of training
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | DSR Ankle | Predicate Ankle
Number analyzed (Participants) | 3 | 3
seconds | 0.31 (0.13) | 0.27 (0.19)

3. Secondary Outcome: Orthotics Prosthetics User Survey (OPUS) Device Satisfaction
Description: The OPUS is a self-report questionnaire consisting of 5 modules. It can be used for prosthetic and orthotic programs for quality assessment, to maintain awareness of improvement in activities, to evaluate changes in patient's functional status and quality of life, and to assess satisfaction with devices and services. The Device Satisfaction module uses a 5-point Likert scale (1 to 5), with a total score range of 11 to 55. Higher values indicate higher levels of satisfaction.
Time Frame: after up to 3 weeks of training
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DSR Ankle | Predicate Ankle
Number analyzed (Participants) | 2 | 2
units on a scale | 45 (5.66) | 44.5 (3.54)

4. Secondary Outcome: 10 Meter Walk Test (10 MWT)
Description: The 10 MWT assesses walking speed in meters per second over a distance of 10 meters.
Time Frame: after up to 3 weeks of training
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | DSR Ankle | Predicate Ankle
Number analyzed (Participants) | 3 | 2
meters per second | 0.41 (0.28) | 0.53 (0.29)

5. Secondary Outcome: Six Minute Walk Test (6 MWT)
Description: The 6 MWT assesses walking distance in meters over a period of 6 minutes.
Time Frame: after up to 3 weeks of training
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | DSR Ankle | Predicate Ankle
Number analyzed (Participants) | 2 | 2
meters | 145.1 (121.48) | 162.9 (142.84)

6. Secondary Outcome: Timed Up and Go (TUG)
Description: The TUG assesses mobility, balance, walking ability, and fall risk in older adults.
Time Frame: after up to 3 weeks of training
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | DSR Ankle | Predicate Ankle
Number analyzed (Participants) | 2 | 2
seconds | 42.17 (26.16) | 23.13 (14.87)

ADVERSE EVENTS:
Time Frame: For each intervention, the period of time for adverse event monitoring was the 3 to 4 hour period during which the device was worn for the in-lab gait sessions. The participants did not wear the experimental intervention for home or daily use in this study.
Description: The risks associated with study participation are no greater than minimal risk as defined in 45 CFR 46.102(i): "Minimal risk means that the probability and magnitude of harm or discomfort anticipated in the research are not greater in and of themselves than those ordinarily encountered in daily life or during the performance of routine physical or psychological examinations or tests."
Arm/Group | DSR Ankle | Predicate Ankle
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT05955378/Prot_SAP_ICF_000.pdf